CLINICAL TRIAL: NCT06954480
Title: An Open-label Randomised, Phase II Trial of Datopotamab Deruxtecan Plus Durvalumab Versus Datopotamab Deruxtecan in Patients With PDL1-negative Metastatic Triple-negative Breast Cancer
Brief Title: Investigating Datopotamab Deruxtecan Plus Durvalumab Versus Datopotamab Deruxtecan in Patients With PDL1-negative Metastatic Triple-negative Breast Cancer
Acronym: DIAMOND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1011098
Record Dates: First submitted 2025-03-14; First posted 2025-05-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; breast cancer; PDL1-negative; Datopotamab Deruxtecan; Durvalumab
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dato-DXd plus Durva (Experimental): In arm A, patients will receive Durvalumab 1120mg plus Dato-DXd 6.0mg/kg.
  Interventions: Drug: Datopotamab Deruxtecan (Dato-DXd); Drug: Durvalumab
- Arm B - Dato-DXd (Active Comparator): In arm B, patients will receive Dato-DXd 6.0mg/kg.
  Interventions: Drug: Datopotamab Deruxtecan (Dato-DXd)

INTERVENTIONS:
Drug: Datopotamab Deruxtecan (Dato-DXd) — Patients will receive Dato-DXd 6.0mg/kg, which will be administered by infusion on day 1 of each 21-day cycle.
Drug: Durvalumab — Patients will receive Durva 1120mg, which will be administered by infusion on day 1 of each 21-day cycle.
  Arms: Dato-DXd plus Durva

SUMMARY:
The DIAMOND study is being carried out to evaluate if Datopotamab deruxtecan (Dato-DX) in combination with Durvalumab is more effective than Dato-DXd alone in treating PDL1-negative advanced or metastatic triple negative breast cancer (TNBC). Globally, breast cancer is the most common malignancy in women and the second most common cancer overall. The term TNBC is used to define tumours that do not express oestrogen receptors, progesterone receptors and HER2 receptors. TNBC comprises 10 -15% of all breast cancers. It remains the subtype with poorest outcome and there is a significant need to develop new therapies for this group of patients especially. Moreover, the PDL1-negative tumour has demonstrated no benefit from standard 1st line treatment of chemotherapy plus immune checkpoint inhibitors.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate the superiority of Datopotamab deruxtecan (Dato-DXd) plus Durvalumab (Durvalumab) relative to Dato-DXd alone in patients with PDL1-negative advanced or metastatic triple negative breast cancer (TNBC). This is also the primary endpoint of this study and effectivenss measured by progression-free survival. Dato-DXd is an antibody drug conjugate (ADC) that targets tumour-associated calcium signal transducer 2, TROP2, a transmembrane protein that is highly expressed in various epithelial tumors including breast cancer. Durvalumab is an immune checkpoint inhibitor and is expected to stimulate the patient's anti-tumour immune response by binding to PD-L1 and shifting the balance toward an anti-tumour response. The preclinical and clinical evidence have suggested synergistic activity between antibody drug conjugate and immune checkpoint inhibitor. This study will recruit 140 patients, aged 18 and over and consenting patients will be randomly placed into one of two treatment groups. One group will receive Datopotamab deruxtecan in combination with Durvalumab and the other groups will receive Datopotamab deruxtecan alone. Treatment will continue unless there is evidence of unacceptable toxicity, disease progression, or if the patient requests to stop the treatment or death. Safety and tolerability as well as progression free survival, overall survival, clinical benefit rate, duration of response and duration of clinical benefit and quality of life will be assessed.

PD-L1 is part of a complex system of receptors and ligands that are involved in controlling T-cell activation. The PD-1 receptor (cluster of differentiation [CD]279) is expressed on the surface of activated T cells. It has 2 known ligands: programmed cell death ligand-1 (PD-L1; B7-H1; CD274) and programmed cell death ligand-2 (PD-L2; B7-DC; CD273). PD-L1/PD-L2 belong to a family of immune checkpoint proteins that act as coinhibitory factors, which can halt or limit the development of T cell response. When PD-L1 binds to PD-1, an inhibitory signal is transmitted into the T cell, which reduces cytokine production and suppresses T cell proliferation. Tumour cells exploit this immune checkpoint pathway as a mechanism to evade detection and inhibit immune response.

Sites will perform local PD-L1 testing to confirm the PD-L1 status of potentially eligible patients. PD-L1 negativity in this trial will be defined as 22C3 Combined Positive Score (CPS) of less than 10.

Durvalumab is a human mAb of the immunoglobulin G (IgG) 1 kappa subclass that blocks the interaction of PD-L1 (but not PD-L2) with PD-1 on T cells and CD80 (B7.1) on immune cells. The proposed mechanism of action for durvalumab is interference in the interaction of PD-L1 with PD-1 and CD80 (B7.1). The blockade of PD-L1/PD-1 and PD-L1/CD80 interactions releases the inhibition of immune responses, including those that may result in tumor elimination. In vitro studies demonstrate that durvalumab antagonizes the inhibitory effect of PD-L1 on primary human T cells, resulting in restored interferon-gamma (IFN-γ)-induced proliferation. In vivo studies have shown that durvalumab inhibits tumor growth in xenograft models via a T cell-dependent mechanism. Based on these data, durvalumab is expected to stimulate the patient's antitumor immune response by binding to PD-L1 and shifting the balance toward an antitumor response. Durvalumab has been engineered to reduce antibody-dependent cellular cytotoxicity and complement-dependent cytotoxicity.

Dato-DXd is an antibody drug conjugate that targets tumour-associated calcium signal transducer 2, TROP2, a transmembrane protein that is highly expressed in various epithelial tumours including breast cancer. TROP2 has several binding partners, including claudin 1, claudin 7, cyclin D1, protein kinase C, phosphatidylinositol 4,5-bisphosphate, and insulin-like growth factor 1. By binding to these targets, TROP2 affects tight junctions at the epithelial barrier and increases tumour proliferation, podosome formation, and Raf and NF-kappa activation and suppresses IGF-1R signaling [21,22]. Its expression correlates with aggressive tumour behaviour and has been used as a prognostic marker in several types of cancer.

DNA topoisomerase I is an enzyme that acts by causing a transient break in 1 strand of DNA. This enables the unwinding of positive or negative supercoiled DNA through a hindered rotary system, thus allowing the separation of the double-helix strands. This activity is prominent during cell replication. Inhibition of DNA topoisomerase I can lead to cell apoptosis following multiple breaks in the cell DNA. DNA topoisomerase I has therefore been identified as a potential target for cancer treatment.

In order to overcome the challenges of delivering cytostatics specifically into cancer cells, ADCs have been developed. ADCs are composed of an antibody, a linker, and a cytotoxic agent. ADCs are payload delivery systems that can target cells that express the preferred marker. The ADC specifically binds and is internalized into the target cells, and enzymatic processes release the drug into the cytoplasm.

Dato-DXd binds to TROP2, is internalized, and undergoes enzymatic processing. Thereafter the DNA Dato-DXd binds to TROP2, and after further enzymatic processing, the DNA topoisomerase I inhibitor DXdis released, inhibits cell replication, and promotes cell apoptosis. The anti-TROP2 component, is a humanized IgG1 kappa monoclonal antibody. The released drug is a DNA topoisomerase I inhibitor derivative of exatecan. The monoclonal antibody is covalently conjugated to a drug-linker, which is composed of a cleavable maleimide tetrapeptide linker and the released drug. The tetrapeptide linker is designed to be stable in plasma to reduce systemic exposure to the released drug.

In vitro studies indicate that Dato-DXd exhibits TROP2 expression-dependent cell growth inhibitory activity, and in vivo studies using a tumor-bearing mouse model indicate that administration of Dato-DXd results in the regression of TROP2-positive tumors. The biodistribution and antitumor activity of the ADC are expected to depend on the expression level of the target antigen in tumor tissue.Dato-DXd has been evaluated in multiple solid tumors ,including NSCLC, and TNBC, HR+/HER2- BC, and urothelial cancer have high expression of TROP2, 1,2 and the DNA topoisomerase I inhibitor, irinotecan, shows clinical efficacy in these indications 9,10. Dato-DXd has shown preliminary efficacy in the ongoing clinical studies.

The screening period for the trial is 28 days. Following randomisation, patients must commence on trial treatment within 3 days.

There are specific protocol mandated pre-randomisation eligibility criteria that needs to be fulfilled, which includes the below:

1. Assessing eligibility thoroughly using the protocol inclusion and exclusion criteria and obtaining informed consent.
2. Conducting local PD-L1 assessment and confirming PD-L1 negativity by 22C3 Combined Positive Score (CPS) of less than 10.
3. A representative formalin-fixed, paraffin embedded (FFPE) tumour specimen with the supporting report is required to enable the definitive diagnosis of TNBC, with adequate viable tumour cells in a tissue block.
4. Obtaining medical history and demographics.
5. Confirming ECOG performance status.
6. Completing limited physical exam (including clinical breast examination), vital sins and weight with height.
7. Haematology and Biochemistry bloods.
8. Urinalysis.
9. Pregnancy test.
10. Thyroid function test.
11. Coagulation and Virology test.
12. Yearly ophthalmologic assessment if done as routine standard of care.
13. CT tumour assessment (using RECIST v1.1).
14. Brain scan.
15. Collection of adverse events and concomitant medications.
16. Completion of QOL questionnaires.
17. Collection if research blood samples.

Once the above assessments have satisfactorily completed, the sponsor team, CECM DIAMOND coordinating team will check the screening eCRF data against the protocol and confirm eligibility. Once this has been completed, site staff can then proceed to randomising the patient on the Interactive Response Technology (IRT) system. Both the site and pharmacy staff and the CECM coordination team will receive a confirmation of randomisation via email.

Patients will be randomised in 1:1 rations to receive one of the two following treatment arms:

1. Dato-DXd (Dose 6mg/kg, IV) plus Durvalumab (1120 mg, IV) on Day 1 Q3W.
2. Dato-DXd (Dose 6mg/kg) on Day 1 Q3W.

Randomisation will be stratified as a three-part stratification by the following:

1. Is de novo; or
2. has treatment-free interval of < = 12 months or
3. has a treatment-free interval of > 12 months

Throughout the duration of the trial treatment, the below assessments will be performed (+/- 3 days) and associated data collected and reported on the eCRF:

1. ECOG performance status.
2. Limited physical exam (including clinical breast examination), vital sins and weight with height.
3. Haematology and Biochemistry bloods.
4. Pregnancy test.
5. Thyroid function test.
6. CT tumour assessment (using RECIST v1.1) every 9 weeks until disease progression.

6. Yearly ophthalmologic assessment if done as routine standard of care. 7. Adverse events and concomitant medications. 8. QOL questionnaires. 9. Patient review for safety occurring only on day 14 from cycle 1 to 3, where information on adverse events on concomitant medications will be collected.

During the safety visit, which occurs 90 days after the last dose (+/- 7 days), the below assessments will be performed and associated data collected and reported on the eCRF:

1. ECOG performance status.
2. Limited physical exam (including clinical breast examination), vital sins and weight with height.
3. Haematology and Biochemistry bloods.
4. Pregnancy test.
5. Thyroid function test.
6. Ophthalmologic assessment if done as routine standard of care.
7. Adverse events and concomitant medications.
8. QOL questionnaires.

Upon disease progression, the below assessments will be performed and associated data collected and reported on the eCRF:

1. CT tumour assessment (using RECIST v1.1).
2. Adverse events and concomitant medications.
3. Optional fresh tumour biopsy.
4. Research blood samples.

When a patient discontinues study treatment, they will be followed up for subsequent anti-cancer therapies, disease and survival status until death, loss to follow-up or withdrawal of consent (whichever comes first) All patients will be followed up for survival until 2 year post last patient treatment discontinuation. Each patient will be followed up at least every 6 months in the follow up period. If patient requests to be withdrawn from follow-up; this request must be documented in the source documents and signed by the investigator. If the patient withdraws from study treatment but not from follow-up, the study staff may use patient medical records to obtain information about subsequent anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol.
3. Female ≥ 18 years of age.
4. Triple-negative disease, defined as tumour cells being:

   * Negative for ER with <10% of tumour cells positive for ER on IHC or IHC score (Allred) of ≤3.
   * Negative for PR with <10% of tumour cells positive for PR on IHC or IHC score (Allred) of ≤3 or PR unknown, and
   * Negative for HER2 with 0, 1+ or 2+ intensity on IHC and no evidence of amplification on ISH.
5. PDL1 negative, defined as 22C3 CPS<10.
6. Patients must have:

   * at least one lesion, not previously irradiated, that can be measured accurately at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computed tomography (CT) or magnetic resonance imaging (MRI) performed within 28 days prior to randomisation which is suitable for accurate repeated measurements, or
   * lytic or mixed (lytic + sclerotic) bone lesions in the absence of measurable disease as defined above; patients with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible. Patient that cannot be assessed by the CT or MRI should be excluded from the study.
7. Representative formalin-fixed paraffin embedded (FFPE) breast tumour samples with an associated pathology report from the primary or recurrent cancer that are determined to be available and sufficient for central testing OR tumour accessible for biopsy.
8. ECOG performance status 0-1.
9. Life expectancy ≥12 weeks.
10. Adequate haematologic and end-organ function within 28 days prior to the first study treatment defined by the following:

    * Absolute neutrophil count ≥ 1500 cells/μL (1.5 x 109/L) (without granulocyte) colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1).
    * WBC > 2500/μL (2.5 x 109/L).
    * Platelet count ≥ 100,000/μL (100 x 109/L) (transfusion not permitted within 28 days of study medication).
    * Haemoglobin ≥ 9.0 g/dL (90g/L) with no blood transfusions (packed red blood cells).
    * Serum albumin ≥ 3g/dL.
    * AST (SGOT) or ALT (SGPT) and ALP ≤ 2.5 times the institutional upper limit of normal (ULN), bilirubin ≤ 1.5 x ULN (patients with liver metastases who have AST or ALT ≤ 5 x the institutional ULN may be enrolled).
    * aPTT ≤ 1.5 × the institutional ULN, INR <1.5 and absence of evidence of impaired hepatic synthesis function. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
    * Serum Creatinine ≤ 1.5 x institutional ULN.
    * Glomerular filtration rate ≥ 40mL/min as assessed by standard methodology at the investigating center (i.e., Cockcroft Gault, MDRD or CKD-EPI formulae, EDTA clearance or 24 h urine collection).
    * No evidence of haematuria: +++ on microscopy or dipstick.
11. Patients of childbearing potential are eligible provided they have a negative serum or urine pregnancy test on Cycle 1, Day 1 (within 72 hours) of study treatment, preferably as close to the first dose as possible. Patients must agree to use adequate contraception, defined as those methods with a failure rate of < 1 % per year beginning 14 days before the first dose of study drug and for 7 months after the last dose of study drug. Also, participants must not donate, or retrieve for their own use, ova at any time during this study and for at least 7 months after the last dose of treatment. Preservation of ova should be considered prior to randomisation or the first dose of study intervention.
12. Body Weight > 30 kg.

Exclusion Criteria:

1. Prior chemotherapy, immunotherapy (including durvalumab) or treatment with PARP inhibitors for advanced or metastatic breast cancer.
2. Prior treatment with immune checkpoint inhibitors (eg atezolizumab, pembrolizumab) or DNA topoisomerase I or TROP2- or HER2-targeting ADCs and TROP2 targeted therapy in the (neo)adjuvant setting within 6 months from the end of treatment and randomisation into this study.
3. Patients with prior allogeneic stem cell or solid organ transplantation.
4. Patients must not have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent), or had oral or IV steroids for 14 days prior to the first dose of study drug; the use of intranasal, inhaled corticosteroids topical steroids, or local steroid injections, physiologic replacement doses of glucocorticoids (i.e. for adrenal insufficiency) and mineralocorticoids (e.g. fludrocortisone) or steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication is allowed.
5. Administration of a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Active or prior documented autoimmune or inflammatory disorders including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, , rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis , Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement therapy
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included
   * Patients with celiac disease controlled by diet alone
7. History of idiopathic pulmonary fibrosis (including pneumonitis or interstitial lung disease), drug-induced pneumonitis, radiation pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia) requiring steroids, or evidence of active pneumonitis on screening chest CT scan.
8. Active infection requiring systemic therapy.
9. History of HIV infection.
10. Known active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
11. Known history of active tuberculosis (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
12. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
13. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the study protocol.
14. Concurrent treatment with other experimental drugs or participation in another clinical trial with therapeutic intent within 28 days prior to randomisation.
15. Pregnant and lactating female patients.
16. Major surgical procedure within 4 weeks prior to randomisation or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
17. Malignancies other than breast cancer within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent).
18. Severe infections within 28 days prior to randomisation in the study including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
19. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

    * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
20. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, situations that would limit compliance with study requirement, substantially increase risk of incurring AEs.
21. History of leptomeningeal carcinomatosis.
22. Has clinically significant corneal disease.
23. Has a history of severe hypersensitivity reactions to other monoclonal antibodies.
24. History of active primary immunodeficiency.
25. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
26. Brain metastases or neoplastic spinal cord compression. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression. In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent and anticonvulsants for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.
27. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
28. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
PFS is defined as the time from the date of randomisation to the date of first documented confirmed tumour progression (using RECIST 1.1) or death from any cause, whichever occurs first in all patients. | PFS is defined as the time from the date of randomisation to date of first documented confirmed disease progression or death, which ever occurs first, assessed on average up to 12 months.
  PFS is defined as the time from randomisation to disease progression or relapse (as assessed by the site radiologist and/or investigator, using RECIST, Version 1.1) or death on study from any cause (defined as death within 30 days of the last study treatment), whichever occurs first. For patients who have not died or experienced disease progression at the end of study, PFS will be censored on the last date the patient was known to be progression free.

SECONDARY OUTCOMES:
OS is defined as the time from date of randomisation to the date of death due to any cause in all patients. | From date of randomisation to the date of death due to any cause in all patients, assessed on average up to 12 months.
  Overall survival is defined as the time from randomisation to death from any cause. All deaths will be included, whether they occur on study or following treatment discontinuation. For patients who have not died, overall survival will be censored at the date of last contact.
DoR is defined as the time from first documentation of CR or PR to confirmed disease progression using RECIST 1.1, or death on study from any cause, whichever occurs first, in patients with objective response. | The time from first documentation of CR or PR to confirmed disease progression, or death on study from any cause, whichever occurs first in patients with objective response, assessed on average up to 12 months.
CBR is defined as the percentage of patients who have achieved at least one CR or PR or met the SD criteria at least once after randomisation for a minimum interval of 24 weeks continuously (using RECIST 1.1). | Up to 24 weeks
  Clinical Benefit rate is defined as number of patients with complete or partial response or stable disease maintained ≥24 weeks (as assessed by the site radiologist and/or investigator, using RECIST1.1) divided by the number of patients in the analysis. Patients without a post-baseline tumour assessment will be considered to have no clinical benefit. An estimate of the clinical benefit rate and 95% CIs (Blyth-Still-Casella; 21-22) will be calculated for each treatment arm. CIs for the difference in clinical benefit rate (Satner and Snell 1980; Berger and Boos 1994; 23-24) will be calculated. The relative risk (treatment:control) will be reported along with the associated 95% confidence interval. Statistical inference will be evaluated using Chi-square statistic; the Fisher's exact test may be used if the expected counts in some cells are small.
DoCB is calculated as time (in months) from randomisation to progression or death from any cause in patients with a clinical benefit. | From the time (in months) from randomisation to progression or death from any cause in patients with a clinical benefit, assessed on average up to 12 months..
  For patients with an objective response, duration of objective response is defined as the time from initial complete or partial response to disease progression or death on study from any cause (defined as death within 30 days of the last study treatment), whichever occurs first. For patients with a clinical benefit (objective response or stable disease maintained ≥24 weeks), duration of clinical benefit is defined as the time from randomisation to disease progression or death on study from any cause (defined as death within 30 days of the last study treatment), whichever occurs first. Methods for handling censoring and for analysis are the same as those described for PFS.
Changes in quality of life measured by the time to deterioration (TTD) | From the time of enrollment to the safety visit (90 days +/- 7 days after the last dose.), assessed up to at least 122 PFS events have occured
  Changes in quality of life measured by the time to deterioration (TTD) in Items 29 (overall health) and 30 (overall QoL) of the EORTC Quality of Life Questionnaire Core 30 (QLQ-C30) and the percentages of patients with a decrease or increase of ≥ 10 points on the global health status/HRQoL scale of the EORTC QLQ-C30 and on subsets, respectively.
  Patient reported outcome assessment is one type of clinical outcome assessment and is a general term referring to all outcomes and symptoms that are directly reported by the participant. PROs have become important in evaluating the efficacy and tolerability of study interventions in clinical studies and will aid in understanding of the benefit/risk evaluation.
Incidence, nature and severity of adverse events with severity determined according to CTCAE v5.0. | From the time of enrollment to the safety visit (90 days +/- 7 days after the last dose.), assessed up to at least 122 PFS events have occurred

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, MD PhD, FRCP, Study Director — Queen Mary University of London
Locations (2):
- United Kingdom (2):
  - Barts Cancer Institute, Centre of Experimental Cancer Medicine, London
  - Barts Health NHS Trust, London